CLINICAL TRIAL: NCT01979315
Title: Cross Correlation of Pain Hypersensitivity and Clinical and EMG Parameters
Brief Title: Cross Correlation of Pain Hypersensitivity and Clinical Features and Electromyography in Low Back Pain Patients
Status: Completed | Type: Observational
Sponsor: University of Belgrade (Other)
Responsible Party: Principal Investigator, Konstantinovic Ljubica, professor, University of Belgrade
Other Study IDs: LK-1
Record Dates: First submitted 2013-10-25; First posted 2013-11-08 (Estimated); Last update posted 2021-11-16 (Actual); Status verified 2021-11

CONDITIONS: Low Back Pain
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 5 Days
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- patients with LBP
- healthy individulas

SUMMARY:
Diagnostic and prognostic value of pain hypersensitivity in low back pain (LBP) is not fully understood.Increased pain sensitivity in the primary area of pain (local pain) is considered a sign of predominantly peripheral pain sensitization,value of pain hypersensitivity in low back pain (LBP)is not fully understood whereas pain sensitivity in distal and remote areas is considered to present a more central phenomenon. It is suggested that pat ents with enhanced pain sensitivity report high level of disability. Despite fact that pain and disability are associated in chronic LBP the exact mechanisms of sensitivity contribution in LBP disability is unknown. It has also been suggested that muscle function changes may be driven by pain. The possible role and contribution of trunk muscles function to pain and disability phenomena remain unknown.

This study was aimed to estimate prevalence and possible correlation among pain hypersensitivity and functional and electromyography parameters of trunk muscles in patients reporting early phase of chronic LBP.

ELIGIBILITY:
Inclusion Criteria:

* Low back pain for at least 12 weeks
* Magnetic resonance imaging (MRI) confirmation of prolapsed intervertebral disc (PID)
* No meeting excluding criteria.

Exclusion Criteria:

* No response to initial contact
* Red flag symptoms
* Diabetes mellitus,
* Neurological problems and
* Cancer
* Pregnant patients
* Patients treated chirurgically for the same problem or treated with oral corticosteroids and steroid injections for any reason in the previous month.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with subacute LBP from tertiary rehabilitation clinic
Sampling Method: Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2015-12 (Actual); Primary Completion 2021-01 (Actual); Study Completion 2021-05 (Actual)

PRIMARY OUTCOMES:
Pain hypersensitivity parameters: pain threshold and pressure pain tolerance threshold will be measured by pressure algometer pressure was applied using a probe with an area of 1 cm2 and intensity to a maximum of 1,000 kPa at a rate of 30 kPa/s. | up to 3 months
  pain detection threshold and pressure pain tolerance threshold (PPTT) )will be measured at the site of maximal pain and of more distant nonpainful point at the back, and the ipsilateral great toe 3 times and average value will be taken for statistics analyses

CONTACTS AND LOCATIONS:
Locations (1):
- Clinic for rehabilitation dr Miroslav Zotovic Faculty of Medicine University of Belgrade, Belgrade, Serbia